CLINICAL TRIAL: NCT00253357
Title: Predictors of Response to Cardiac Re-Synchronization Therapy
Brief Title: PROSPECT: Predictors of Response to Cardiac Re-Synchronization Therapy
Status: Completed | Type: Observational
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Collaborators: Medtronic (Industry)
Other Study IDs: 226
Record Dates: First submitted 2005-11-13; First posted 2005-11-15 (Estimated); Last update posted 2007-12-21 (Estimated); Status verified 2007-12

CONDITIONS: Heart Failure; Congestive Heart Failure; Cardiomyopathy
Keywords: Heart Failure; Congestive Heart Failure; Fluid overload; Left sided heart failure; Pacemaker; Defibrillator
MeSH Terms: conditions — Heart Failure; Cardiomyopathies; Edema

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Heart failure is a progressive disease that decreases the pumping action of the heart. This may cause a backup of fluid in the heart and may result in heart beat changes. Using a medical device like a pacemaker or a defibrillator can help the heart to pump in regular beats. However, not all patients do better with a device. Currently, there is not a way to identify which patients will benefit from the device. The purpose of this study is to determine if using medical tests, Echocardiogram, can help in predicting which patients will improve. The types of patients needed for this study are those who have been diagnosed with moderate or severe heart failure.

ELIGIBILITY:
Inclusion Criteria:

* Moderate to severe heart failure

  * Ejection Fraction ( measurement of blood pumped out of the heart) less than 35%
  * Wide (greater than 130 milliseconds) QRS duration for US patients only.
  * May include patients with less than 130 millisecond QRS duration if they have mechanical dyssynochrony (uncoordinated heart contractions) in Europe.
  * All patients enrolled should be stable on medications that include at least an ACE inhibitor or Angiotensin Receptor Blocker (ARB) and at optimal level for at least one month prior to surgery

Exclusion Criteria:

* Patients that are not eligible for this study are those that have a mechanical right heart valve or are experiencing the following medical conditions within the last 3 months:

  * Chest pain / unstable angina
  * Acute heart attack
  * Chronic or permanent atrial arrhythmias such as atrial fibrillation
  * Contrary artery bypass graft (CABG)
  * Percutaneous transluminal coronary angioplasty (PTCA)
  * Patients who have had intermittent or continuous Inotropic drug therapy are not eligible for this study.
  * Patients who have had heart transplant or a prior Cardiac Resynchronization Therapy device are not eligible for this study.
  * Patients who are pregnant or are of child-bearing potential are not on a form of birth control may not participate in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450
Dates: Start 2004-03; Study Completion 2006-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William T Abraham, MD, Principal Investigator — University of Ohio
Locations (28):
- United States (16):
  - Several Locations, California
  - Gainsville, Florida
  - Atlanta, Georgia
  - Columbus, Illinois
  - Kansas City, Kansas
  - New Orleans, Louisiana
  - Grand Rapids, Michigan
  - Several Locations, New Jersey
  - Several Locations, New York
  - Winston-Salem, North Carolina
  - Several Locations, Ohio
  - Dolyestown, Pennsylvania
  - Nashville, Tennessee
  - Burlington, Vermont
  - Norfolk, Virginia
  - Seattle, Washington
- Several Locations, Austria
- Several Locations, Belgium
- Several Locations, Denmark
- Several Locations, Finland
- Several Locations, France
- Several Locations, Germany
- Several Locations, Hong Kong
- Several Locations, Italy
- Several Locations, Netherlands
- Several Locations, Norway
- Several Locations, Spain
- Several Locations, United Kingdom

REFERENCES:
- [Derived] Hsing JM, Selzman KA, Leclercq C, Pires LA, McLaughlin MG, McRae SE, Peterson BJ, Zimetbaum PJ. Paced left ventricular QRS width and ECG parameters predict outcomes after cardiac resynchronization therapy: PROSPECT-ECG substudy. Circ Arrhythm Electrophysiol. 2011 Dec;4(6):851-7. doi: 10.1161/CIRCEP.111.962605. Epub 2011 Sep 28. PMID 21956038
- [Derived] Chan PS, Khumri T, Chung ES, Ghio S, Reid KJ, Gerritse B, Nallamothu BK, Spertus JA. Echocardiographic dyssynchrony and health status outcomes from cardiac resynchronization therapy: insights from the PROSPECT trial. JACC Cardiovasc Imaging. 2010 May;3(5):451-60. doi: 10.1016/j.jcmg.2009.08.012. PMID 20466340
- [Derived] Chung ES, Leon AR, Tavazzi L, Sun JP, Nihoyannopoulos P, Merlino J, Abraham WT, Ghio S, Leclercq C, Bax JJ, Yu CM, Gorcsan J 3rd, St John Sutton M, De Sutter J, Murillo J. Results of the Predictors of Response to CRT (PROSPECT) trial. Circulation. 2008 May 20;117(20):2608-16. doi: 10.1161/CIRCULATIONAHA.107.743120. Epub 2008 May 5. PMID 18458170